CLINICAL TRIAL: NCT05626309
Title: Qizhu Yuling Prescription in the Prevention and Treatment of Postoperative Metastasis and Recurrence of Esophagus Cancer：A Randomized, Double-blind, Controlled and Multi-center Clinical Study
Brief Title: Clinical Trial of Qizhu Yuling Prescription in the Prevention and Treatment of Esophagus Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jie Li (Other)
Responsible Party: Sponsor-Investigator, Jie Li, Vice President, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Organization: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-1-4151
Record Dates: First submitted 2022-10-31; First posted 2022-11-23 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Esophagus Cancer
Keywords: Postoperative esophagus cancer; Qizhu Yuling prescription; Chinese Herbal Medicine; Randomized Controlled Trial; 1-year disease-free survival rate
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qizhu Yuling Prescription (Experimental): Qizhu Yuling Prescription
  Interventions: Drug: Qizhu Yuling Prescription
- Placebo Comparator (Placebo Comparator): Simulation agent of Qizhu Yuling Prescription Group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Qizhu Yuling Prescription — The dosage form of the test drug is granule. Patients need to take 2 small packets in the morning and 2 small packets in the evening. The medicine needs to be melted in hot water before being taken. Every 4 weeks is a course of treatment, a total of 6 courses,The patients were followed up to 3 years after esophageal cancer surgery.
  Arms: Qizhu Yuling Prescription
Drug: Placebo — It is prepared from maltodextrin and food coloring. The raw materials of maltodextrin conform to the relevant provisions of excipients - maltodextrin in the fourth part of Chinese Pharmacopoeia 2015 edition. Food coloring includes caramel coloring, egg yolk coloring and milk chocolate brown pigment, all of which are edible grade ingredients. Patients need to take 2 small packets in the morning and 2 small packets in the evening. The medicine needs to be melted in hot water before being taken. Every 4 weeks is a course of treatment, a total of 6 courses,The patients were followed up to 3 years after esophageal cancer surgery.
  Other Names: Simulation agent of Qizhu Yuling Prescription
  Arms: Placebo Comparator

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Qizhu Yuling prescription for postoperative esophagus cancer.

DETAILED DESCRIPTION:
This study include a multi-center, randomized, double-blind, placebo, parallel controlled clinical trial.The randomized clinical trial will enroll approximately 310 patients. Participants will be randomly divided into experimental (n=155) and placebo groups (n=155).Patients in the experimental group was treated with Qizhu Yuling prescription within 6 months after esophagus cancer R0. Patients in the control group will receive the placebo.The primary endpoint is 1-year DFS (Disease-free survival) rate after surgery, that refers to the proportion of patients who do not have recurrence, metastasis or death (from any cause) within 1 years after surgery. The research protocol was approved by the relevant ethics committees, and the study was conducted according to the Declaration of Helsinki and Good Clinical Practice guidelines. Patients gave written informed consent to participate in the trial.

ELIGIBILITY:
Inclusion Criteria:

* 1. Esophageal cancer without esophagogastric junction pT1-4aN + M0 (stage IIB-IVA) meeting the diagnostic criteria without recurrence or metastasis;

  2. Patients who have completed adjuvant therapy (including adjuvant radiotherapy, adjuvant chemotherapy, adjuvant chemotherapy + radiotherapy) within 6 months after R0 resection for esophageal cancer;

  3. ECOG score 0-2;

  4. 18-75 years old;

  5. Expected survival ≥ 3 months;

  6. Subjects voluntarily signed informed consent.

Exclusion Criteria:

* 1. Combined with primary tumor at other sites;

  2. Patients complicated with severe primary diseases of heart, cerebral vessels, liver, kidney and hematopoietic system;

  3. Patients with mental illness and mental and language disorders;

  4. Participation in other clinical trials within 3 months;

  5. Patients with known hypersensitivity or intolerance to study drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
1-year disease-free survival rate | The day of surgery until the first year
  Refers to the proportion of patients who did not experience recurrence, metastasis or death (from any cause) within 1 years after surgery.

SECONDARY OUTCOMES:
Disease-free survival | Randomization until disease recurrence, metastasis, death (from any cause) , or 36 months after surgery, whichever occurs first.
  It is the time from randomization to tumor progression or death (from any cause).
Overall survival | Randomization until death (from any cause) or 36 months after surgery, whichever occurs first.
  It is the time from randomization to death (from any cause).
Cumulative annual recurrence and metastasis rate for 1-3 years | The day of surgery until the once, second and third year.
  Refers to the proportion of patients with recurrence and metastasis within 1-3 years from the day of surgery.
Cumulative annual survival rate for 1-3 years | The day of surgery until the once, second and third year.
  Refers to the proportion of patients with survical within 1-3 years from the day of surgery.
Indexes related to fat distribution | before and after every third cycles of treatment (each cycle is 28 days), assessed up to recurrence and metastasis (up to 3 years after surgery).
  Total Fat Area, Visceral Fat Area and Subcutaneous Fat Area. They measure fat area on cross-sectional images using plain CT scanning.
Visceral Adiposity Index | before and after every third cycles of treatment (each cycle is 28 days), assessed up to recurrence and metastasis (up to 3 years after surgery).
  It is a new assessment of visceral fat based on waist circumference (WC), BMI, triglyceride (TG) and HDL.
  Male VAI = during [WC/(39.68 + 1.88 x BMI)] * (TG / 1.03) * (1.31 / HDL). Female VAI = during [WC/(36.58 + 1.89 x BMI)] * (TG / 0.81) * (1.52 / HDL).
Tumor marker | before and after every third cycles of treatment (each cycle is 28 days), assessed up to recurrence and metastasis (up to 3 years after surgery).
  CEA
Tumor marker | before and after every third cycles of treatment (each cycle is 28 days), assessed up to recurrence and metastasis (up to 3 years after surgery).
  SCC
Tumor marker | before and after every third cycles of treatment (each cycle is 28 days), assessed up to recurrence and metastasis (up to 3 years after surgery).
  CYFR21-1
Tumor marker | before and after every third cycles of treatment (each cycle is 28 days), assessed up to recurrence and metastasis (up to 3 years after surgery).
  CA199
Peripheral blood inflammatory index LMR | before and after every third cycles of treatment (each cycle is 28 days), assessed up to recurrence and metastasis (up to 3 years after surgery).
  The ratio of lymphocytes to monocytes (LMR)
Peripheral blood inflammatory index LNR | before and after every third cycles of treatment (each cycle is 28 days), assessed up to recurrence and metastasis (up to 3 years after surgery).
  The ratio of Lymphocyte to neutrophil ratio (LNR)
Prognostic nutritional index | before and after every third cycles of treatment (each cycle is 28 days), assessed up to recurrence and metastasis (up to 3 years after surgery).
  Serum albumin level (g/L) +5× total number of peripheral blood lymphocytes (×10 ^ 9 /L)
Quality of life of the patient (QLQ-QES18) | Before and after every cycle of treatment (each cycle is 28 days), assessed up to death or 3 years after surgery.
  The score will be measured by Quality of Life Questionnaire of Oesophageal-Specific Module 18. Each question is scored from 1 to 4 with 18 questions giving a total score of 18 to 72. A higher score indicates a poorer quality of life.
Evaluation of the patient's symptoms (MDASI-TCM) | Before and after every cycle of treatment (each cycle is 28 days), assessed up to death or 3 years after surgery.
  The score will be measured with M. D. Anderson Symptom Traditional Chinese Medicine. Each question is scored from 0 to 10 with 26 questions for a total score of 0 to 260. A higher score indicates a poorer symptom.
Medication compliance | From randomization to the end of the sixth course of medication （up to 24 weeks）.
  The number of cases and percentage were calculated as < 80%, 80-120% and > 120%
Percentage of Participants With Adverse Events | aseline until disease progression, death, or assessed up to 36 months after surgery.
  Percentage of Participants With Adverse Events in different arms.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Li, Professor, Study Director — Guang 'anmen Hospital, China Academy of Chinese Medical Sciences; Yu Wu, Professor, Principal Investigator — Xiyuan Hospital of China Academy of Chinese Medical Sciences; Shijie Zhu, Professor, Principal Investigator — Wangjing Hospital, China Academy of Chinese Medical Sciences; Guowang Yang, Professor, Principal Investigator — Beijing Hospital of Traditional Chinese Medicine
Locations (3):
- China (3):
  - Beijing Hospital of Traditional Chinese Medicine, Capital Medical University, Beijing, Beijing Municipality
  - Xiyuan Hospital, China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality
  - Wangjing Hospital, China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Yes
The results of the study will be issued to publications through scientific journals and conference reports. The anonymized datasets used and/or analyzed during the current study are available from the sponsor-investigator on reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Kong M, Xu B, Zhu G, Wang X, Kuang Z, Sun Q, Liu K, Wang Z, Zhang Y, Li J. Qizhu Yuling prescription in the prevention of postoperative metastasis and recurrence of esophagus cancer: study protocol for a randomized, double-blind, placebo-controlled, multicenter clinical trial. Front Oncol. 2025 Mar 26;15:1478390. doi: 10.3389/fonc.2025.1478390. eCollection 2025. PMID 40206581